CLINICAL TRIAL: NCT04038203
Title: Resonance Raman Spectroscopy Detects Peripheral Tissue Oxygen Deprivation in Very Low Birth Weight Infants With Umbilical Artery Catheters
Brief Title: Tissue Oxygen Deprivation as Detected With Raman in Association With Umbilical Artery Catheters
Status: Withdrawn | Type: Observational
Why Stopped: IRB expired. The Study will not be resumed.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201900739; OCR25462 (Other: UF OnCore)
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Tissue Oxygenation
Keywords: neonates; low birth weight; spectroscopy; Umbilical Artery Catheter (UAC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates with UAC placement: Neonates with birth weight less than 1500 grams with UAC placed on admission. Raman measurements will be obtained simultaneously on the right AND left lower extremity for 15 minutes daily in the first week of life.
  Interventions: Device: Resonance Raman Spectroscopy (RPS)

INTERVENTIONS:
Device: Resonance Raman Spectroscopy (RPS) — RRS is a technology that utilizes vibrational spectroscopy, rather than absorbance spectroscopy, to determine the oxyhemoglobin concentration in tissues. Raman measurements for the UAC neonates will be obtained simultaneously on the right AND left lower extremity for 15 minutes daily in the first week of life.
  Other Names: Raman

SUMMARY:
Umbilical artery catheters (UACs) are associated with significant morbidity in preterm neonates however are necessary for the management of this high risk population. UACs have been linked to serious adverse events (SAEs) including arterial thrombosis, necrotizing enterocolitis, limb ischemia, and renal failure. Resonance Raman Spectroscopy (RRS), raman for short, is a technology that utilizes vibrational spectroscopy, rather than absorbance spectroscopy, to determine the oxyhemoglobin concentration in tissues.

In this prospective, observational study, daily measurements of StO2 of low birth weight neonates using raman spectroscopy will be correlated with UACs.The study team hypothesizes that raman can detect changes in peripheral tissue oxygenation in the ipsilateral extremity to the UAC and that raman is more sensitive at detecting changes in peripheral tissue oxygenation then common metrics used to monitor neonatal hemodynamics. If successful, this study would demonstrate that raman can be used as an early marker of tissue oxygen deprivation in neonates with UACs and maybe used to guide management in other clinical scenarios where StO2 is affected.

ELIGIBILITY:
Inclusion Criteria:

* Neonate Inclusion Criteria:

  1. Birth weight less than 1500 grams.
  2. Admitted to the NICU.
  3. UAC placed on admission.
* Mother Inclusion Criteria:

  1. Admitted to the labor and delivery or antenatal floors with reasonable chance of delivery of a neonate weighing less than 1500 grams as determined by the obstetrics team.

Exclusion Criteria:

* Neonate Exclusion Criteria:

  1. Neonates with congenital heart defects or major congenital anomalies such as known or suspected inborn errors of metabolism, ambiguous genitalia, neural tube defects, malignancy, abdominal wall defects, airway defects and chromosomal anomalies.
* Mother Exclusion Criteria:

  1. Mother is pregnant with fetus with congenital heart defect or major congenital anomaly as described above.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonates with birth weight less than 1500 grams, admitted to the University of Florida neonatal intensive care unit (NICU), with UAC placed on admission.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a Significant Adverse Event (SAEs) | Week 1
  SAEs will be a composite of any of the following: lower extremity ischemia, Acute Kidney Injury (AKI), Neo natal Necrotizing Enterocolitis (NEC) or death abstracted from the medical record and/or bedside nurse interview, if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Ruoss, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Children's Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shahid S, Dutta S, Symington A, Shivananda S; McMaster University NICU. Standardizing umbilical catheter usage in preterm infants. Pediatrics. 2014 Jun;133(6):e1742-52. doi: 10.1542/peds.2013-1373. Epub 2014 May 19. PMID 24843063
- [Background] Elboraee MS, Toye J, Ye XY, Shah PS, Aziz K; Canadian Neonatal Network Investigators. Association between Umbilical Catheters and Neonatal Outcomes in Extremely Preterm Infants. Am J Perinatol. 2018 Feb;35(3):233-241. doi: 10.1055/s-0037-1606607. Epub 2017 Sep 14. PMID 28910847
- [Background] McAdams RM, Winter VT, McCurnin DC, Coalson JJ. Complications of umbilical artery catheterization in a model of extreme prematurity. J Perinatol. 2009 Oct;29(10):685-92. doi: 10.1038/jp.2009.73. Epub 2009 Jun 25. PMID 19554012
- [Background] Huxtable RF, Proctor KG, Beran AV. Effect of umbilical artery catheters on blood flow and oxygen supply to extremities. Pediatr Res. 1976 Jul;10(7):656-60. doi: 10.1203/00006450-197607000-00005. PMID 934731
- [Background] Iyengar A, Gaillardetz A, Tighiouart H, Castillo B, Romfh P, Davis JM. Direct Measurement of Tissue Oxygenation in Neonates via Resonance Raman Spectroscopy: A Pilot Study. Neonatology. 2017;112(2):137-142. doi: 10.1159/000458514. Epub 2017 May 18. PMID 28514777
- [Background] Lin SJ, Koltz PF, Davis W, Vicari F. Lower extremity ischemia following umbilical artery catheterization: a case study and clinical update. Int J Surg. 2009 Jun;7(3):182-6. doi: 10.1016/j.ijsu.2008.12.038. Epub 2008 Dec 25. PMID 19349222
- [Background] Ward KR, Barbee RW, Reynolds PS, Torres Filho IP, Tiba MH, Torres L, Pittman RN, Terner J. Oxygenation monitoring of tissue vasculature by resonance Raman spectroscopy. Anal Chem. 2007 Feb 15;79(4):1514-8. doi: 10.1021/ac061072x. PMID 17297949
- [Background] Robert B. Resonance Raman spectroscopy. Photosynth Res. 2009 Aug-Sep;101(2-3):147-55. doi: 10.1007/s11120-009-9440-4. Epub 2009 Jul 1. PMID 19568956
- [Background] Spiro TG. Resonance Raman spectroscopy as a probe of heme protein structure and dynamics. Adv Protein Chem. 1985;37:111-59. doi: 10.1016/s0065-3233(08)60064-9. PMID 2998161
- [Background] Gay AN, Lazar DA, Stoll B, Naik-Mathuria B, Mushin OP, Rodriguez MA, Burrin DG, Olutoye OO. Near-infrared spectroscopy measurement of abdominal tissue oxygenation is a useful indicator of intestinal blood flow and necrotizing enterocolitis in premature piglets. J Pediatr Surg. 2011 Jun;46(6):1034-40. doi: 10.1016/j.jpedsurg.2011.03.025. PMID 21683194
- [Background] Gordon PV, Swanson JR, Attridge JT, Clark R. Emerging trends in acquired neonatal intestinal disease: is it time to abandon Bell's criteria? J Perinatol. 2007 Nov;27(11):661-71. doi: 10.1038/sj.jp.7211782. Epub 2007 Jul 5. PMID 17611610